CLINICAL TRIAL: NCT04912024
Title: Comparative Outcome Measures of Patients Receiving Acute Renal ThErapy Study (COMPARE)
Brief Title: Comparative Outcome Measures of Patients Receiving Acute Renal ThErapy Study
Acronym: COMPARE
Status: Completed | Type: Observational
Sponsor: Outset Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-04
Record Dates: First submitted 2021-05-26; First posted 2021-06-03 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: End Stage Kidney Disease; End Stage Renal Disease; Acute Kidney Injury
Keywords: Tablo; Outset Medical; ESRD; AKI
MeSH Terms: conditions — Kidney Failure, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Tablo Hemodialysis System: Participants who were prescribed acute intermittent renal replacement therapy on the Tablo Hemodialysis System at a dialysate flow rate of 300 mL/min
  Interventions: Device: Intermittent Renal Replacement Therapy using the Tablo Hemodialysis System
- Conventional Hemodialysis System: Participants who were prescribed acute intermittent renal replacement therapy on conventional hemodialysis systems (Non-Tablo) with dialysate flow rates of ≥ 500 mL/min
  Interventions: Device: Intermittent Renal Replacement Therapy using Conventional Hemodialysis Systems

INTERVENTIONS:
Device: Intermittent Renal Replacement Therapy using the Tablo Hemodialysis System — Intermittent renal replacement therapy using the Tablo Hemodialysis System in the acute setting for participants with AKI or ESKD
  Groups: Tablo Hemodialysis System
Device: Intermittent Renal Replacement Therapy using Conventional Hemodialysis Systems — Intermittent renal replacement therapy using Conventional Hemodialysis Systems in the acute setting for participants with AKI or ESKD
  Groups: Conventional Hemodialysis System

SUMMARY:
Retrospective, multicenter, comparative, post-market study of the Tablo Hemodialysis System in hospitalized participants with End-Stage Renal Disease or Acute Kidney Injury.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age.
* Participant weighs ≥ 34kg.
* Participant was hospitalized and had dialysis dependent End-Stage Renal Disease or Acute Kidney Injury and was prescribed acute intermittent renal replacement therapy.

Exclusion Criteria:

* Treatments isolated to ultrafiltration only.
* Any documented condition the Physician feels would prevent the participant from successful inclusion in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with AKI or ESKD who were prescribed acute intermittent Renal Replacement Therapy (RRT).
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
BUN Lab Value | Change from baseline BUN measurement at 24 hours.
  Change in Blood Urea Nitrogen

SECONDARY OUTCOMES:
Bicarbonate Lab Value | Change from baseline bicarbonate measurement at 24 hours.
  Change in Bicarbonate
Potassium Lab Value | Change from baseline potassium measurement at 24 hours
  Change in Potassium

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Adventist Health System, Orlando, Florida
  - Texas Health Harris Methodist Hospital Fort Worth, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.